CLINICAL TRIAL: NCT03893370
Title: A Sham Controlled Prospective Randomized Clinical Trial of the RejuvenAir® System for the Treatment of Moderate to Severe Chronic Obstructive Pulmonary Disease With Chronic Bronchitis
Brief Title: RejuvenAir® System Trial for COPD With Chronic Bronchitis
Acronym: SPRAY-CB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 016
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Chronic Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic

STUDY DESIGN:
Intervention Model Description: randomized, sham-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Treatment (Active Comparator): RJA MCS
  Interventions: Device: RejuvenAir System
- Sham Control (Sham Comparator): Sham
  Interventions: Device: Sham Control Procedure

INTERVENTIONS:
Device: RejuvenAir System — RejuvenAir Metered CryoSpray
  Arms: Treatment
Device: Sham Control Procedure — Sham Control Procedure
  Arms: Sham Control

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is defined as an impaired ability to move air within the lungs and is a major public health problem that is projected to rank fifth worldwide in terms of disease burden and third in terms of mortality. Chronic bronchitis (CB) is a common clinical phenotype within the umbrella of a COPD diagnosis and is classically defined as chronic cough and sputum production for 3 months a year for 2 consecutive years2, but many studies have used different definitions to define it- chronic cough and sputum production for one year or cough and sputum production on most days of the week. CB is associated with multiple clinical consequences, including; the worsening of lung function decline, increasing risk of acute exacerbations of COPD, increased risk of developing pneumonia, reduced health related quality of life, and an increase in all-cause mortality.

DETAILED DESCRIPTION:
The RejuvenAir® System is a cryosurgical device that applies medical-grade liquid nitrogen to the treatment area via a radial head catheter in a small, accurately directed spray. Cryotherapy with the RejuvenAir® System is designed to induce a regenerative endobronchial tissue effect by: 1) destroying via cryotherapy the abnormal surface epithelium that has become overgrown with mucin producing goblet cells, 2) thus allowing normal bronchial epithelium with a regrowth of ciliated epithelial cells that will facilitate the removal of mucins from the bronchial airways and 3) lead to a reduction in chronic inflammation and its accompanying mucosal swelling with resultant increase in the treated airway diameter. This reversal of inflamed epithelium may also lessen systemic inflammation.

ELIGIBILITY:
Inclusion Criteria

* Males and females ≥40 to ≤80 years of age
* Subject is able to read, understand, and sign a written Informed Consent in order to participate in the Study
* Subject has a diagnosis of chronic bronchitis (CB) and/or chronic obstructive pulmonary disease (COPD) for a minimum of two years. (Chronic Bronchitis is defined clinically as chronic productive cough for 3 months in each of 2 successive years in a patient in whom other causes of productive cough have been excluded)
* Subject is classified as having a moderate or severe (GOLD 2/3) airflow obstruction defined by a post-bronchodilator of ≥30% FEV1 to <80% predicted with a baseline FEV1/FVC of <0.70
* Subject has a Baseline SGRQ of ≥50
* Subject demonstrates daily cough and significant mucus.
* Subject is being treated according to current medically accepted treatment guidelines for chronic bronchitis for minimum of 3 months prior to enrollment into the study. Subject agrees to continue maintenance pulmonary/COPD medications (GOLD standard medications recommended) for the duration of the study
* Non-smoking for a minimum of 2 months prior to consent and agrees to continue not smoking for the duration of the study
* Subject is able to adhere to and undergo 2 bronchoscopic procedures (cross over subjects may undergo two additional bronchoscopic procedures, if they agree to treatment), per hospital guidelines
* Subject demonstrates ability and willingness to use a daily eDiary

Exclusion Criteria

* Subject has had an acute pulmonary infection, exacerbation or pneumonia requiring medical treatment (with antibiotics and/or steroids) within 4 weeks prior of initially planned study bronchoscopy
* Current diagnosis of Asthma
* Subject has Alpha-1 antitrypsin deficiency as defined by blood level <59 mg/dL
* Subject has other origins of respiratory disease aside from chronic bronchitis and COPD
* Subject is using e-cigarettes, vaping or taking any inhaled substances not prescribed by a physician
* Subject has untreatable or life threatening arrhythmias, inability to adequately oxygenate during the bronchoscopy, or has acute respiratory failure
* Subject has bullous emphysema characterized as large bullae >30 millimeters on HRCT; or subject has stenosis in the tracheobronchial system, tracheobronchomegaly, trachea-bronchomalacia, amyloidosis or cystic fibrosis
* Subject has clinically significant bronchiectasis
* Subject has had a solid transplant procedure
* Subject has a known mucosal tear, has undergone prior lung surgery such as pneumonectomy, lobectomy, bullectomy, or lung volume reduction surgery
* Subject has had a prior lung device procedure, including emphysema stent(s) implanted, lung coils, valves, lung denervation, bronchial thermoplasty, cryotherapy or other therapies
* Subject is unable to temporarily discontinue use of anticoagulant therapy: warfarin, Coumadin, LMWH, heparin, clopidrogel (or equal)
* Subject has a serious medical condition, such as: uncontrolled coagulopathy or bleeding disorder, congestive heart failure, uncontrolled angina, myocardial infarction in the past year, renal failure, liver disease, cerebrovascular accident within the past 6 months, uncontrolled diabetes, uncontrolled hypertension or uncontrolled gastric reflux
* Subject is pregnant, nursing, or planning to get pregnant during study duration
* Subject has or is receiving chemotherapy or active radiation therapy within the past 6 months or is expected to receive chemotherapy during participation in this study
* Subject is or has been in another treatment study within 6 weeks of enrollment and agrees to not participate in any other treatment studies for the duration of study participation
* Subject has known sensitivity to medication required to perform bronchoscopy (such as lidocaine, atropine, and benzodiazepines)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire | 12 months
  Change in St. George Respiratory Questionnaire (SGRQ) score from Baseline to 12 months

SECONDARY OUTCOMES:
Subjects experiencing serious adverse events (SAEs) rated as probably or definitely related to the study device or procedure | Within 30 days after either the first or second study procedure
  Number of subjects experiencing one or more serious adverse events (SAEs) rated as probably or definitely related to the study device or procedure by the investigator within 30 days after either the first or second study procedure.
Reduction of cough | Baseline through 12 months
  Reduction of cough from Baseline through 12 months
Reduction of sputum | Baseline through 12 months
  Reduction of sputum from Baseline through 12 months
Acute Exacerbation Rate (AECOPD) | 12 months
  Acute Exacerbation rate (AECOPD, all severities) over 12 months
COPD assessment test (CAT) score | 12 months
  COPD assessment test (CAT) from Baseline through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University Health System
Locations (27):
- United States (26):
  - Honor Health, Scottsdale, Arizona
  - El Camino Hospital, Mountain View, California
  - University of California, Davis Medical Center, Sacramento, California
  - Advanced Pulmonary Research Institute, Loxahatchee Groves, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Northwestern University, Chicago, Illinois
  - Louisiana State University Medical Center, Shreveport, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins Universtiy, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health, Grand Rapids, Michigan
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Health System, Camden, New Jersey
  - Duke University, Durham, North Carolina
  - University Of Cincinnati, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State Universisty, Columbus, Ohio
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - Temple University - Of the Commonwealth System of Higher Education, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health - Midlands, Columbia, South Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - St. David's Georgetown Hospital, Georgetown, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No